CLINICAL TRIAL: NCT00616005
Title: Phase II Treatment of Adults With Primary Malignant Glioma With Irinotecan Plus Temozolomide
Brief Title: Ph. II Treatment of Adults w Primary Malignant Glioma w Irinotecan + Temozolomide
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00012939; 8044 (Other: DUMC)
Record Dates: First submitted 2008-02-03; First posted 2008-02-14 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2010-08

CONDITIONS: Glioblastoma
Keywords: Glioblastoma; GBM; Brain tumor; Temodar; Temozolomide; Irinotecan; CPT-11; Camptosar; Malignant glioma; Anaplastic astrocytoma; Glioblastoma multiforme
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms; Glioma; Astrocytoma | interventions — Temozolomide; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Other): Pts taking EIAEDs
  Interventions: Drug: Temodar and Irinotecan
- 2 (Other): Pts not taking EIAEDs
  Interventions: Drug: Temodar and Irinotecan

INTERVENTIONS:
Drug: Temodar and Irinotecan — Temozolomide-orally 200mg/m2 in fasting state 1hr prior to CPT-11 infusion. Temozolomide-day 1 of treatment cycle & every 24hrs thereafter for 5days w treatment cycles repeated every 6wks. Treatment cycles repeated up to maxi of 3 cycles until occurrence of either unacceptable toxicity/evidence of disease progression. CPT-11-intravenously in fasting state over 90min. CPT-11 1hr after Temozolomide administration on day 1 of treatment cycle. CPT-11-days 1, 8, 22, & 29 of 6wk treatment cycle. Treatment cycles may be repeated up to maxi of 3 cycles until occurrence of either unacceptable toxicity/evidence of disease progression. Dose of CPT-11 will be based on whether pt is receiving EIAEDs due to increased drug clearance produced by agents. For pts receiving EIAEDs, CPT-11 dose of 325mg/m2 administered. For pts not receiving EIAEDs, CPT-11 dose of 125mg/m2 administered.
  Other Names: Temodar - Temozolomide; Irinotecan - Camptosar - CPT11

SUMMARY:
Objective:

To determine activity of combo of Irinotecan + Temozolomide To further characterize any toxicity associated w combo of Irinotecan + Temozolomide

DETAILED DESCRIPTION:
Objectives of study are to determine activity of combo of Irinotecan + Temozolomide & to further characterize any toxicity associated w combo of Irinotecan + Temozolomide. Temozolomide administered orally at 200mg/m2 in fasting state 1hr prior to CPT-11 infusion. Temozolomide administered on day 1 of treatment cycle & every 24hrs thereafter for 5 days w treatment cycles repeated every 6wks. Treatment cycles may be repeated up to maxi of 3 cycles until occurrence of either unacceptable toxicity/evidence of disease progression. At end of 3rd cycle/if cycles are stopped early for toxicity or progression, subject will undergo radiation therapy. CPT-11 administered intravenously in fasting state over 90min. CPT-11 will begin 1hr after Temozolomide administration on day 1 of treatment cycle. CPT-11 administered on days 1, 8, 22, & 29 of 6wk treatment cycle. Treatment cycles may be repeated up to maxi of 3 cycles until occurrence of either unacceptable toxicity/evidence of disease progression. Dose of CPT-11 will be based on whether pt is receiving CYP3A4-inducing antiepileptic drugs due to increased drug clearance produced by these agents. For pts receiving EIAEDs including phenytoin, fosphenytoin, oxcarbazepine, phenobarbital/ primidone, CPT-11 dose of 325mg/m2 administered. For pts not receiving EIAEDs, CPT-11 dose of125 mg/m2 administered.

Subjects have newly diagnosed histologically proven supratentorial glioblastoma multiforme. Toxicities associated w CPT-11 are anemia, decreased blood counts, diarrhea, constipation, nausea, vomiting, tiredness, fever, mouth sores, dehydration, rash, itching, changes in skin color, swelling, numbness, tingling, dizziness, confusion, low blood pressure, sweating, hot flashes, hair loss, inflammation of liver, flu-like symptoms, decreased urine output, shortness of breath,& pneumonia. Low white blood cell & platelet counts may be associated w risk of infection/bleeding, respectively. Irinotecan has also caused birth defects in animals. Most frequent toxicities in earlier studies have been low white blood cells & diarrhea, & death has been seen from these & other side effects. Temozolomide has been well tolerated by both adults & children w most common toxicity being mild myelosuppression. Other, less likely, potential toxicities include nausea & vomiting, constipation, headache, alopecia, rash, burning sensation of skin, esophagitis, pain, diarrhea, lethargy, hepatotoxicity, anorexia, fatigue & hyperglycemia. Hypersensitivity reactions have not yet been noted w Temozolomide. As in case w many anti-cancer drugs, Temozolomide may be carcinogenic.

ELIGIBILITY:
Inclusion Criteria:

* Pts have histologically proven supratentorial GBM
* Pts have newly diagnosed disease
* There must be measurable disease on contrast-enhanced magnetic resonance imaging performed <14 days before drug administration. Those who underwent resection must have MRI <72 hrs/ >14 days after surgery
* Prior Surgical Resection/Biopsy: Although surgical resection is not required, pts must be treated <42 days of surgery or biopsy
* Age >18 yrs
* Karnofsky Performance Status >70 percent
* Serum creatinine < 1.5 x ULN
* Absolute neutrophil count >1500 cells/microliter; platelet count >100,000 cells/microliter
* Serum SGOT & total bilirubin <2.5 x ULN
* Signed informed consent, approved by IRB, will be obtained prior to initiating treatment
* Pts must agree to practice effective birth control measures while on study & for 2 months after completing therapy

Exclusion Criteria:

* Pregnant/breast feeding women / women/men w reproductive potential not practicing adequate contraception. This therapy may be associated w potential toxicity to fetus/child that exceeds minimum risks necessary to meet health needs of mother
* Active infection requiring intravenous antibiotics
* Known diagnosis of HIV infection
* Pts w history of another primary malignancy that currently requires active intervention
* Pts unwilling/unable to comply w protocol due to serious medical/psychiatric condition
* Pts who underwent surgical resection for GBM <2 weeks of start of treatment
* Pts who have received prior chemo, biologic therapy, XRT, interstitial brachytherapy/radiosurgery to brain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2005-11; Primary Completion 2007-07 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 6 months

SECONDARY OUTCOMES:
Toxicity assessment | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: David A. Reardon, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

REFERENCES:
- See also: The Preston Robert Tisch Brain Tumor Center at DUKE — http://www.cancer.duke.edu/btc/